CLINICAL TRIAL: NCT02881307
Title: Ultrasound Assessment of Rheumatoid Arthritis Patients Who Changed Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veena Ranganath, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Veena Ranganath, MD, MS, Associate Clinical Professor, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Weight Loss Ultrasound RA Proj
Record Dates: First submitted 2016-08-19; First posted 2016-08-26 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Overweight
Keywords: Rheumatoid Arthritis (RA); Musculoskeletal Ultrasound (MSUS)
MeSH Terms: conditions — Arthritis, Rheumatoid; Overweight | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Ultrasonographer and joint assessor are blinded to the diet intervention and to each others assessments.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement (Experimental)
  Interventions: Dietary Supplement: Whey Protein&Prebiotic Supplement; Behavioral: Dietary recommendations
- Dietary Counseling (Active Comparator)
  Interventions: Behavioral: Dietary Counseling

INTERVENTIONS:
Dietary Supplement: Whey Protein&Prebiotic Supplement — Dietary supplement (protein drink) commercially available protein shakes
  Arms: Dietary Supplement
Behavioral: Dietary Counseling — Dietary Counseling
  Arms: Dietary Counseling
Behavioral: Dietary recommendations — recommendations for one meal per day including lean protein and vegetables
  Arms: Dietary Supplement

SUMMARY:
The purpose of this research study is to evaluate if a weight loss intervention will improve your rheumatoid arthritis disease activity.

DETAILED DESCRIPTION:
This is a pilot 12-week RCT (Randomized Clinical Trial) in 60 obese RA (Rheumatoid Arthritis) patients to evaluate if a weight loss intervention will improve PDUS (Power Doppler Ultra Sound), traditional disease activity measures (DAS28, Disease Activity Score - 28), and adipokine/MBDA (Multi-Biomarker Disease Activity) assessments. While there have been observational weight loss RA studies, none were RCTs and they did not utilize objective measures (PDUS or MBDA).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must meet 1987 ACR (American College of Rheumatology) criteria
2. Age > 18 years of age
3. Baseline DAS28/ESR>3.2 (ESR-erythrocyte sedimentation rate)
4. Stable DMARDs or biologic therapy for at least 12 weeks, or stable off RA therapy 12 weeks.
5. Willingness to participate in a weight loss program
6. BMI > 30
7. Prednisone ≤ 10 mg
8. Patient has provided informed consent

Exclusion Criteria:

1. Major surgery (including joint surgery) within 8 weeks prior to baseline or planned major surgery within 3 months after baseline
2. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease
3. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (as this may falsely elevate biomarkers)
4. Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of baseline or oral antibiotics within 2 weeks prior to baseline
5. Pregnant women or nursing (breast feeding) mothers
6. Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation
7. History of an eating disorder
8. History of bariatric surgery
9. EKG results deeming patient to unsafe for study intervention
10. Allergy to study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
change in PDUS | change from baseline to 6 and 12 months
  Change in Synovitis measure using Ultrasound
change in DAS28 | change from baseline to 6 and 12 months
  Change in DAS28 represents conventional measure of reduced disease activity

SECONDARY OUTCOMES:
MBDA | Baseline, 6 weeks and 12 weeks
  Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Veena K Ranganath, M.D., M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ranganath VK, La Cava A, Vangala S, Brook J, Kermani TA, Furst DE, Taylor M, Kaeley GS, Carpenter C, Elashoff DA, Li Z. Improved outcomes in rheumatoid arthritis with obesity after a weight loss intervention: randomized trial. Rheumatology (Oxford). 2023 Feb 1;62(2):565-574. doi: 10.1093/rheumatology/keac307. PMID 35640116